CLINICAL TRIAL: NCT06382571
Title: Factors Associated With Sub - Targeted Therapeutic Dose Of Renin - Angiotensin Blockage Among Chronic Heart Failure With Reduced Ejection Fraction Patients
Status: Completed | Type: Observational
Sponsor: Chulalongkorn University (Other)
Responsible Party: Sponsor
Other Study IDs: 026/66
Record Dates: First submitted 2024-02-20; First posted 2024-04-24 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-02

CONDITIONS: Heart Failure With Reduced Ejection Fraction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Sub - target dose group: Patients who received sub - target dose of Angiotensin converting enzyme inhibitors (ACEIs), angiotensin receptor-neprilysin inhibitors (ARNIs), and angiotensin receptor blockers (ARBs).
  Interventions: Drug: Renin-Angiotensin System Inhibitor
- Target dose group: Patients who received target dose or maximal tolerated dose of Angiotensin converting enzyme inhibitors (ACEIs), angiotensin receptor-neprilysin inhibitors (ARNIs), and angiotensin receptor blockers (ARBs)
  Interventions: Drug: Renin-Angiotensin System Inhibitor

INTERVENTIONS:
Drug: Renin-Angiotensin System Inhibitor

SUMMARY:
Objective: To analyze factors associated with Thai heart failure with reduced ejection fraction patients who received sub-target doses of Angiotensin converting enzyme inhibitors (ACEIs), angiotensin receptor-neprilysin inhibitors (ARNIs), and angiotensin receptor blockers (ARBs).

Methods: The retrospective cohort study was designed to collect data on Thai heart failure with reduced ejection fraction patients at Out-patient Clinic, Trat Hospital and Phrapokklao Hospital from January 2016 to December 2020. Thirteen factors were analyzed to determine their association with the sub-target group.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were first diagnosed be heart failure with left ventricular ejection fraction less than 40%.
* Received one of ACEIs,ARBs,ARNI drugs.

Exclusion Criteria:

* Electronic medical records was not complete enough to analyse.
* Patients who had history of heart transplantation or had heart transplantation plan in last 12 months.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult out - patients who were first diagnosed be heart failure with left vetricular ejection fraction less than 40% and recieved one of ACEIs,ARBs,ARNI drugs.
Sampling Method: Non-Probability Sample
Enrollment: 396 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
factors associated with sub - target dose of ACEIs,ARBs,ARNI | 12 months
  factors associated with Thai heart failure with reduced ejection fraction patients who received sub-target doses of Angiotensin converting enzyme inhibitors (ACEIs), angiotensin receptor-neprilysin inhibitors (ARNIs), and angiotensin receptor blockers (ARBs).